CLINICAL TRIAL: NCT06284551
Title: The Relationship Between Internet-use Behavior and Mental Health in Youth
Status: Enrolling by invitation | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202111069RINB
Record Dates: First submitted 2024-02-15; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Mental Health Issue
Keywords: youth; cyberbullying; mental health; social media addiction; internet gaming disorder; suicide/self-injury; depression; anxiety; emotional regulation
MeSH Terms: conditions — Cyberbullying; Psychological Well-Being; Internet Addiction Disorder; Depression; Anxiety Disorders; Emotional Regulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Healthy youths and adults aged 15-24 years old.
- Experimental Group: Youths and adults aged 15-24 years old with diagnosis of major depressive disorder, anxiety disorder, post traumatic stress disorder, or Adjustment disorder according to DSM-V.

SUMMARY:
Introduction: WHO defines youth as 15-24 years age group. At this stage, the brain is still under development, with high impulsiveness, being fond of stimulation and yearning for peer life. Compared with traditional interpersonal interaction, modern youths use the Internet as a main interpersonal interaction platform and conduct lots of leisure activities on the Internet. Poor cognitive emotion regulation strategies and personal traits may extend to new types of mental health issues; and are associated with depression, anxiety, suicidal/self-injurious behaviors, and cyberbullying.

Objectives: (1) To investigate whether emotion regulation strategies while facing stressful events are highly related to with cyberbullying, social media, and internet gaming disorder. (2) To investigate the relation between cyberbullying and depression, anxiety, suicide/self-injury among Taiwanese youths. (3) To investigate the probability of cyberbullying, social media addiction, and internet gaming disorder occurring at the same time.

Method: This cross-sectional study recruits cases of youths from 15 to 24 years old and collects data through questionnaires survey. In addition to collection of basic data, Internet using habits, and medical history, self-rated questionnaires include Suicide/Self-Injury Ideation Questionnaire, The Beck Depression Inventory 2nd Edition, Multidimensional Anxiety Scale for Children-Taiwan version, Cognitive Emotion Regulation Questionnaire, Cyberbullying Questionnaire, and Internet Gaming Disorder Scale-Short Form.

ELIGIBILITY:
Inclusion Criteria:

Control group

* Able to understand the content of all questionnaires
* Healthy youths aged 15-20 years old and adults aged 20-24 years old

Experimental group

* Able to understand the content of all questionnaires
* Youths aged 15-20 years old and adults aged 20-24 years old
* Diagnosed with major depressive disorder, anxiety disorder, post traumatic stress disorder, or Adjustment disorder according to DSM-V

Exclusion Criteria:

* Illiterate or unable to understand the content of the questionnaires
* Diagnosed with organic brain injury, schizophrenia, or bipolar disorder according to DSM-V

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Aged from 15 to 24 years old. Healthy youths and adults recruited publicly. Patients with major depressive disorder, anxiety disorder, post traumatic stress disorder, or Adjustment disorder according to DSM-V recruited from outpatient clinic, emergency ward and day care ward of psychiatry department in National Taiwan University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2025-01-27 (Estimated)

PRIMARY OUTCOMES:
Cyberbullying Questionnaire | Up to 8 weeks
  Suppose the subject was the victimization/perpetrators of cyber-bullying or in the past 2 months, and the cyber-bullying-related experience and feeling in school. The main results were qualitative descriptions and would not apply to statistical analysis.

SECONDARY OUTCOMES:
Beck's Depression Inventory (BDI-II) | Up to 2 weeks
  The BDI-II is a 21-item self-report measure that taps major depression symptoms according to diagnostic criteria listed in the Diagnostic and Statistical Manual for Mental Disorders. Items are summed to create a total score, with higher scores indicating higher levels of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-ting Ko, MS, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No